CLINICAL TRIAL: NCT05889208
Title: Prophylactic Permanent Pacemaker in Patients With Right Bundle Branch Block Undergoing Transcatheter Aortic Valve Implantation
Acronym: TAVI-PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Ashkan Eftekhari, Consultant ass. professor MD PhD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAVI-PACE
Record Dates: First submitted 2023-05-26; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Aortic Stenosis; Right Bundle-Branch Block
Keywords: Trans-catheter aortic valve implantation; Pacemaker
MeSH Terms: conditions — Aortic Valve Stenosis; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic pacemaker implantation (Active Comparator): Brady-pacemaker implantation prior the TAVI-procedure. Pacemaker modus is according to local conditions.
  Interventions: Device: Prophylactic pacemaker implantation
- Usual care (No Intervention): Pacemaker implantation after TAVI if atrioventricular block occurs.

INTERVENTIONS:
Device: Prophylactic pacemaker implantation — Pacemaker implantation prior the TAVI-procedure
  Arms: Prophylactic pacemaker implantation

SUMMARY:
The goal of this clinical trial is to learn about the safety and outcome of prophylactic pacemaker implantation in patients with right bundle-branch block undergoing trans-catheter aortic valve (TAVI) implantation in patients with severe aortic stenosis and left ventricular ejection fraction.Participants will be randomized to:

* Prophylactic pacemaker implantation prior TAVI
* Conservative strategy

DETAILED DESCRIPTION:
BACKGROUND Transcatheter aortic valve implantation (TAVI) is standard of care treatment for patients with severe aortic stenosis ≥ 75 years and/or not eligible for surgical aortic valve replacement 1. There are two types of prosthetic valves: balloon expandable (BE) and self-expandable (SE) types with their distinct features 2. The TAVI-procedure and preexisting conditions in this population entails a risk of permanent pacemaker implantation following TAVI due to conduction disturbances related to the valve implantation and valve type (BE vs. SE). The rate of permanent pacemaker implantation after TAVI is between 2.3 - 36 % depending on valve type and pre-existing conditions3. Major risk factors are right bundle branch block (RBBB), left ventricular outflow track calcification, deeper valve implantation, and SE valves4. Pre-existing RBBB in patients undergoing TAVI occurs in 10% of the cases and it is associated with poor outcome5 in terms of higher pacemaker rate and mortality. Advanced conduction disturbances in patients with pre-existing RBBB occur within three days after the TAVI-procedure6. Hence, pre-existing RBBB is a major risk factor in the TAVI-population with higher mortality7 and needs special attention in peri-operative care. Current European Society Cardiology guidelines do not recommend prophylactic pacemaker implantation in patients without indication for permanent pacing8. However, cardiac pacing is associated with a risk of complications and development of heart failure9, and there is no randomized trial demonstrating a benefit of prophylactic pacemaker implantation in patients with pre-existing RBBB. Although previous observational data suggest prophylactic pacemaker implantation in patients with pre-existing RBBB shortens the TAVI procedure and prevents rehospitalization due to heart block10. Hence, there is a gap in knowledge regarding the outcome of prophylactic permanent pacemaker implantation in patients undergoing TAVI with pre-procedural RBBB and additional risk factors for need of post-procedural permanent pacing. This study aims to evaluate the clinical outcome and safety of prophylactic pacemaker implantation in this high-risk patient group versus a conservative strategy in a randomized clinical trial.

PURPOSE To evaluate safety and outcomes of prophylactic permanent pacemaker implantation in patients with RBBB undergoing TAVI.

HYPOTHESIS Prophylactic permanent pacemaker implantation reduces composite primary outcome in patients with RBBB undergoing TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TAVI indicated by severe valvular aortic stenosis
* Written informed consent
* Left ventricular ejection fraction ≥ 40 %
* Persistent RBBB in 12-lead electrocardiogram (RSR' pattern in V1-3, QRS duration > 120 milliseconds, and wide S wave in leads I, aVL, V5-6)

Exclusion Criteria:

* Other indications for pacemaker implantation or previously implanted pacemaker
* Life expectancy < 1 year
* No written informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Events in the control arm | 12 months
  Composite of all-cause mortality, unplanned pacemaker implantation and new onset of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Eftekhari, Principal Investigator — Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Suh SH, Oh TR, Choi HS, Yang EM, Kim CS, Bae EH, Ma SK, Oh KH, Hyun YY, Sung S, Kim SW; Korean Cohort Study for Outcomes in Patients with Chronic Kidney Disease (KNOW-CKD) Investigators. Bone Mineral Density and All-Cause Mortality in Patients with Nondialysis Chronic Kidney Disease: Results from KNOW-CKD Study. J Clin Med. 2023 Feb 25;12(5):1850. doi: 10.3390/jcm12051850. PMID 36902637
- [Background] van Rosendael PJ, Delgado V, Bax JJ. Pacemaker implantation rate after transcatheter aortic valve implantation with early and new-generation devices: a systematic review. Eur Heart J. 2018 Jun 1;39(21):2003-2013. doi: 10.1093/eurheartj/ehx785. PMID 29420704
- [Background] Maeno Y, Abramowitz Y, Kawamori H, Kazuno Y, Kubo S, Takahashi N, Mangat G, Okuyama K, Kashif M, Chakravarty T, Nakamura M, Cheng W, Friedman J, Berman D, Makkar RR, Jilaihawi H. A Highly Predictive Risk Model for Pacemaker Implantation After TAVR. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt A):1139-1147. doi: 10.1016/j.jcmg.2016.11.020. Epub 2017 Apr 12. PMID 28412434
- [Background] Auffret V, Webb JG, Eltchaninoff H, Munoz-Garcia AJ, Himbert D, Tamburino C, Nombela-Franco L, Nietlispach F, Moris C, Ruel M, Dager AE, Serra V, Cheema AN, Amat-Santos IJ, de Brito FS Jr, Lemos PA, Abizaid A, Sarmento-Leite R, Dumont E, Barbanti M, Durand E, Alonso Briales JH, Vahanian A, Bouleti C, Imme S, Maisano F, Del Valle R, Benitez LM, Garcia Del Blanco B, Puri R, Philippon F, Urena M, Rodes-Cabau J. Clinical Impact of Baseline Right Bundle Branch Block in Patients Undergoing Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2017 Aug 14;10(15):1564-1574. doi: 10.1016/j.jcin.2017.05.030. Epub 2017 Jul 19. PMID 28734885
- [Background] Watanabe Y, Kozuma K, Hioki H, Kawashima H, Nara Y, Kataoka A, Nagura F, Nakashima M, Shirai S, Tada N, Araki M, Takagi K, Yamanaka F, Yamamoto M, Hayashida K. Pre-Existing Right Bundle Branch Block Increases Risk for Death After Transcatheter Aortic Valve Replacement With a Balloon-Expandable Valve. JACC Cardiovasc Interv. 2016 Nov 14;9(21):2210-2216. doi: 10.1016/j.jcin.2016.08.035. PMID 27832846
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Nielsen JC, Andersen HR, Thomsen PE, Thuesen L, Mortensen PT, Vesterlund T, Pedersen AK. Heart failure and echocardiographic changes during long-term follow-up of patients with sick sinus syndrome randomized to single-chamber atrial or ventricular pacing. Circulation. 1998 Mar 17;97(10):987-95. doi: 10.1161/01.cir.97.10.987. PMID 9529267
- [Background] Okuno T, Asami M, Heg D, Lanz J, Praz F, Hagemeyer D, Brugger N, Grani C, Huber A, Spirito A, Raber L, Stortecky S, Windecker S, Pilgrim T. Impact of Left Ventricular Outflow Tract Calcification on Procedural Outcomes After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2020 Aug 10;13(15):1789-1799. doi: 10.1016/j.jcin.2020.04.015. PMID 32763071
- [Background] Bisson A, Bodin A, Herbert J, Lacour T, Saint Etienne C, Pierre B, Clementy N, Deharo P, Babuty D, Fauchier L. Pacemaker Implantation After Balloon- or Self-Expandable Transcatheter Aortic Valve Replacement in Patients With Aortic Stenosis. J Am Heart Assoc. 2020 May 5;9(9):e015896. doi: 10.1161/JAHA.120.015896. Epub 2020 May 2. PMID 32362220